CLINICAL TRIAL: NCT04121117
Title: Usefulness of the Chronic Obstructive Pulmonary Disease-population (COPD-PS) Questionnaire and the COPD-6 Device in the Chronic Obstructive Pulmonary Disease Detection in a Tobacco Detoxication Consultation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-COP6-2018-01
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD; Chronic obstructive pulmonary disease population questionnaire; COPD-PS; COPD-6
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tobacco detoxication cohort: Patients appointed in a tobacco detoxication consultation
  Interventions: Other: Chronic obstructive pulmonary disease screening

INTERVENTIONS:
Other: Chronic obstructive pulmonary disease screening — To verify the tobacco withdrawal, the patients will make a cooximetry.
  For the detection of a possible obstructive pattern a measurement of the ventilatory capacity will be make using the COPD-6 device and for the confirmation of COPD diagnosis and the assesment of the airflow obstruction severity a spirometry will be make.
  The patients will also complete the COPD-PS questionnaire.

SUMMARY:
The aim of this study is to evaluate the usefulness of the chronic obstructive pulmonary disease-population questionnaire (COPD-PS) and the COPD-6 device in the early detection of chronic obstructive pulmonary disease in smoker patients .

ELIGIBILITY:
Inclusion Criteria:

* > 35 years old
* Accumulative tobacco rate > 10 paq-year that go to the tobacco detoxication consultation

Exclusion Criteria:

* Unable to fulfill the questionnarie
* Unable to adequately perform the COPD-6 or forced spirometry maneuvers included in the study.
* Reject to participate and sign the informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smoker patients that are treated in the tobacco detoxication consultation
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the usefulness in the COPD early detection of the combination of the COPD-PS questionnaire and the COPD-6 device. | Up to 12 months after the first consultation
  Verify if the combination of the COPDS-questionnaire (made of different items that allow the detection of chronic airflow obstruction) and the COPD-6 device (tool that measures the ventilatory capacity) is suitable for the COPD early detection.

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Valido Morales, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain